CLINICAL TRIAL: NCT02185443
Title: Stereotactic Body Radiation Therapy for the Treatment of Unresectable Liver Metastases in Patients With Colorectal Adenocarcinoma, Carcinoma of the Anal Canal and Gastrointestinal Neuroendocrine Tumors
Brief Title: Stereotactic Body Radiation Therapy (SBRT) for Unresectable Liver Metastases
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Principal Investigator, Andre Tsin Chih Chen, MD, PhD, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RT-01/2014
Record Dates: First submitted 2014-07-04; First posted 2014-07-09 (Estimated); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Liver Metastases; Colorectal Cancer; Anal Canal Cancer; Gastrointestinal Neuroendocrine Tumors
Keywords: SBRT; radiation; Neoplasm Metastasis; Colorectal Neoplasms; Anal Canal; Neuroendocrine Tumors
MeSH Terms: conditions — Colorectal Neoplasms; Anal Canal Carcinoma; Neoplasm Metastasis; Neuroendocrine Tumors | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SBRT (Experimental)
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: SBRT — * 60Gy in 3 fractions (20Gy/fraction) over 14 days
  * 60Gy in 5 fractions (12Gy/fraction) over 18 days if organ at risk constraints cannot be met with fractionation above
  Other Names: Stereotactic Body Radiation Therapy

SUMMARY:
This is a Phase II study to determine the efficacy of SBRT to treat liver metastases in patients with Colorectal Adenocarcinoma, Carcinoma of the Anal Canal and Gastrointestinal Neuroendocrine Tumors that are not amenable to surgery. Patients should have no evidence of extra-hepatic disease or have disease that is planned to be treated with curative intent.

Therefore, SBRT is being considered as a potentially curative procedure.

ELIGIBILITY:
Inclusion Criteria:

* Karnofsky Performance Scale (KPS) equal or greater than 70
* 1 to 4 liver metastases with an individual maximum diameter of up to 5 cm
* Lesions considered unresectable or patients considered unfit for surgery
* Histology of the primary tumor: colorectal adenocarcinoma, carcinoma of the anal canal or gastrointestinal neuroendocrine tumors.
* Absence of evidence of extra-hepatic disease or extra-hepatic disease to be treated with curative intent.
* Minimum interval of 2 weeks between systemic chemotherapy and SBRT.
* Adequate bone marrow function defined as:
* absolute neutrophils count > 1,800 cells / mm 3
* platelets > 100,000 cells / mm 3
* hemoglobin > 8.0 g / dl ( transfusion or other intervention accepted)

Exclusion Criteria:

* Concomitant chemotherapy
* Prior radiotherapy to the upper abdomen
* Pregnancy
* Underlying Cirrhosis
* Active hepatitis or clinically significant liver failure
* Prior invasive neoplasm except for non-melanoma skin cancer, or unless more than five years without evidence of disease
* Severe Comorbidity
* Current anticoagulant treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2014-05; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Local Progression Free Survival | 2 years
  - Local Progression Free Survival of treated lesions in evaluable patients. Local Progression Free Survival will be defined by the Response Evaluation Criteria in Solid Tumors (RECIST) criteria applied to the Planning Target Volume (PTV) and 1cm around (assessment of marginal failure).
  Time-to-events will be counted from the date of initiation of treatment. Patients will be considered evaluable if followed for at least 6 months after SBRT. A review after 6 months is due to the transient changes after irradiation that make uncertain radiological evaluation before 6 months.

SECONDARY OUTCOMES:
Overall Survival | 5 years
Progression Free Survival | 5 years
Toxicity | 5 years
  treatment related toxicity evaluated by the Common Toxicity Criteria for Adverse Effects (CTCAE) v. 4

CONTACTS AND LOCATIONS:
Overall Officials: Andre TC Chen, MD, PhD, Principal Investigator — Instituto do Cancer do Estado de Sao Paulo
Locations (1):
- Instituto do Cancer do Estado de São Paulo, São Paulo, São Paulo, Brazil